CLINICAL TRIAL: NCT04741568
Title: Development and Feasibility of a Parent Intervention to Prevent Disordered Eating in Children and Young People With Type 1 Diabetes
Brief Title: Parent Intervention to Prevent Disordered Eating in Children With Type 1 Diabetes
Acronym: PRIORITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPON/2020/07/FHMS; 19/0006123 (Other Grant/Funding Number: DiabetesUK)
Record Dates: First submitted 2021-01-15; First posted 2021-02-05 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 1; Disordered Eating; Children, Only; Eating Disorders; Parents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental Psychoeducational Intervention (Experimental): A brief (one-day or two half days) psychoeducation workshop will be provided alongside a website with downloadable content will be made available to review and refresh any skills and techniques. The psychoeducational intervention will be delivered by a research fellow and research assistant with a background in psychology and delivered in line with a protocol.
  Interventions: Behavioral: Parental psychoeducational Intervention
- Wait List Control (No Intervention): Parents randomised to the control arm will be put on the waiting list (wait-list controls) to receive the group intervention after the active treatment group have completed their final follow-up at 3 months.

INTERVENTIONS:
Behavioral: Parental psychoeducational Intervention — The psychoeducation intervention for parents will focus on providing skills, knowledge and support motivation for caregivers of children with diabetes.
  A brief (one-day or two half days) workshop, and a website with downloadable content will be made available to review and refresh any skills and techniques.
  Arms: Parental Psychoeducational Intervention

SUMMARY:
A recent Diabetes UK Position Statement identified several key gaps in the evidence base that might improve mental wellbeing for people with diabetes; one of which was supporting people with diabetes and eating disorders. There is evidence indicating that disordered eating may be more prevalent in children and young people (CYP). Additionally, there is mounting supporting evidence for family-based treatments in both anorexia and bulimia. This study proposes to develop a psycho-education intervention for parents of CYP with Type 1 diabetes (T1D), which will include a one-day workshop with online, downloadable content, and to assess the feasibility of this intervention. Parents will be asked to complete questionnaires about eating habits, diabetes management (both behaviour and knowledge) and wellbeing at three time-points (baseline, one-month and three-months postintervention). Children will also be asked to complete measures on diabetes eating problems at the same time intervals. Parents randomised to the intervention arm will be invited to take part in a semi-structured interview and all parents will be invited to feedback on their participation. It is hypothesised that a psycho-education intervention aimed at parents will help prevent disordered eating in CYP with T1D and improve parental wellbeing.

DETAILED DESCRIPTION:
A recent Diabetes UK Position Statement identified several key gaps in the evidence base that might help improve mental wellbeing for people with diabetes, one of which was supporting people with diabetes and eating disorders. The position statement recommends focusing on people in general, citing studies which observe that 30% of women with T1D omit insulin to control their weight. However, there is evidence indicating that disordered eating may be more prevalent in CYP. A recent meta-analysis found that clinical eating disorders (i.e. anorexia and bulimia) and maladaptive eating and dieting practices (fasting, binge eating, self-induced vomiting, abuse of laxatives, diet pills or other medications including intentional insulin omission - diabulimia) were more prevalent in CYP with T1D (7.0% and 39.3% respectively) than those without T1D (2.7% and 32.5%).

Management of T1D places an inherent focus on dietary intake, specifically carbohydrate counting, physical activity, regular blood sugar monitoring and correct and timely administration of insulin based on these factors. Many high carbohydrate foods can be perceived as 'bad' for blood glucose levels and are subsequently avoided or prohibited within families. This can lead to tensions between CYP and their parents, where CYP may be chastised for eating particular foods or for eating 'forbidden' foods in secret. Additionally, treatment and avoidance of hypoglycaemic episodes can add further complexities to a CYP with T1D's relationship with food, as they may overeat during hypos or save restricted or forbidden foods for hypo treatment. Some CYP may also be discouraged from participating in sport activities due to concerns about a potential hypoglycaemic event. Additionally, depending on age and pre-diagnosis symptoms of T1D, some CYP may also have experienced significant weight loss pre-diagnosis that was quickly regained upon starting insulin treatment; this may provide evidence to CYP that insulin causes them to gain unwanted body weight.

Whilst systematic reviews and meta-analyses exist on the prevalence of eating problems and diabetes as well as associations between eating problems and glycaemic control, the focus of interventions for CYP with T1D has been on the improvement of psychological distress and long-term glycaemic control. Although some interventions included in these reviews have focused on family therapy, they did not explicitly target disordered eating and none were based in the UK. More recently published parenting interventions also do not address disordered eating. Therefore, due to this paucity of evidence for existing interventions, the evidence-base for interventions for clinical eating disorders not specific to T1D is reviewed instead.

The rationale for focusing on interventions aimed at parents is that parents are more responsive to psychological interventions than their offspring. Furthermore, studies have highlighted the protective influence of parents for CYP with clinical eating disorders with family-based treatments playing a key role in supporting CYP in their recovery. Families are a resource in the treatment of eating disorders in CYP and there is mounting evidence that supports family-based treatments in both anorexia and bulimia. Mobilisation of the family system as a resource and an emphasis on promoting specific change early on in treatment in eating disorder-related behaviours have been found to be key elements. The involvement of parents is a key recommendation in the NICE guidelines for eating disorders. Additionally, the Access and Waiting Times Standard for CYP with eating disorders emphasises the necessity of rapid and effective treatment for CYP, along with their families and carers.

Parent-focused psychoeducation groups can be a useful tool to support early change in the treatment of eating disorders. A parent-focused psychoeducation group has been developed at a specialist CYP Eating Disorder service with the aim of offering treatment within a timely manner that promoted early change. The programme is based on key principles from the parenting programme literature and the evidence base for the treatment of eating disorders. Emerging evidence from this group indicated significant positive effects and highlighted that parents benefitted most from the information about managing their CYP's eating disorder and meeting other parents. Another recent evaluation found the group to be an effective source of support for parents, improved their confidence and knowledge in managing their child's eating disorder and their ability to manage their child's adherence to meal plans.

Therefore, it is evident that the involvement of parents could be crucial to facilitate recovery in CYP with eating disorders. Less specific to eating disorders, a recent review of parental interventions to prevent body dissatisfaction or eating disorders in CYP also found encouraging results.

ELIGIBILITY:
Inclusion Criteria:

* Parent or primary caregiver of a CYP aged between 11-14 years with a diagnosis of T1D
* Willing to attend group intervention and provide consent
* Fluent in English or Welsh

Exclusion Criteria:

* Parent receiving psychological support for their child's diabetes and disordered eating
* Parent diagnosis of severe mental health or learning difficulty
* Participating in another trial
* Unable to speak or understand English or Welsh

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Eating Problem Survey Revised (Markowitz et al., 2010) | Baseline, 1-month and 3-months
  A child and parent reported survey of eating problems. Responses are scored on a 6-point Likert scale and higher scores indicate greater eating disorder pathology.

SECONDARY OUTCOMES:
Change in child HbA1c | Baseline, 1-month and 3-months
  Parent reported HbA1c of children
Change in Body Mass Index (weight and height will be combined to report BMI in kg/m^2) | Baseline, 1-month and 3-months
  Parent reported weight and height of children used to calculate BMI
Change in Problem Areas in Diabetes Survey Parent Revised (Markowitz et al., 2012) | Baseline, 1-month and 3-months
  A parent-reported survey to assess diabetes related distress, higher scores indicate greater diabetes distress.
Change in Warwick Edinburgh Mental Wellbeing Scale (Tennant et al., 2007) | Baseline, 1-month and 3-months
  A self report survey to assess parental mental wellbeing. Scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.
Change in Psychological Determinants | Baseline, 1-month and 3-months
  Information Motivation Behvaioural Skills model questionnaire devised for this study completed by parents
Intervention Feedback Survey | 3 months
  Satisfaction and experience with intervention survey devised for this study
Change in Children's Eating Behaviour Questionnaire (Wardle et al. 2001) | Baseline, 1-month and 3-months
  A parent rated instrument to assess eight dimensions of eating style in children. Includes 35 items rates on a 5-point scale, higher scores indicate greater child behaviour for each dimension (e.g. emotional overeating, enjoyment of food).

OTHER OUTCOMES:
Demographics | Baseline
  Parent completed T1D clinical characteristics and healthcare utilisation survey devised for this study (child age, gender, years with diagnosis, number of hospital visits in the last year)
Feasibility Outcomes: Number of Participants Invited to the Study | 3 months
  Number of parents invited to the study
Feasibility Outcomes: Number of Participants Interested in Participating in the Study | 3 months
  Number of Participants Interested in Participating in the Study
Feasibility Outcomes: Number of parents meeting eligibility criteria | 3 months
  Number of parents meeting eligibility criteria
Feasibility Outcomes: Number of parents recruited and participating in the intervention | 3 months
  Number of parents recruited and participate in the intervention
Feasibility Outcomes: Completion Rates (will be calculated from number of parents recruited, number of parents completing the intervention) | 3 months
  We look at the number of enrolled parents who have completed the intervention divided by the total number of parents who have completed the intervention or withdrawn or cancelled.
Feasibility Outcomes: Retention Rates (will be calculated from number of parents recruited and participating in the intervention) | 3 months
  The total number of parents students (including any who have withdrawn), minus the number of parents who have withdrawn or cancelled their enrollment, and divide this by the total number of enrolled parents.
Feasibility Outcomes: Usability of Online Content (Google Analytics) | 3 months
  Analysis on usability of online content. Data obtained from Google Analytics (e.g. website traffic, session duration, pages per session)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jones, PhD, Principal Investigator — University of Surrey
Locations (3):
- United Kingdom (3):
  - Royal Alexandra Children's Hospital, Brighton
  - Royal Surrey Hospital, Guildford
  - Betsi Cadwaladr University Health Board, Holywell

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wylie TAF, Shah C, Connor R, Farmer AJ, Ismail K, Millar B, Morris A, Reynolds RM, Robertson E, Swindell R, Warren E, Holt RIG. Transforming mental well-being for people with diabetes: research recommendations from Diabetes UK's 2019 Diabetes and Mental Well-Being Workshop. Diabet Med. 2019 Dec;36(12):1532-1538. doi: 10.1111/dme.14048. Epub 2019 Jun 19. PMID 31177573
- [Background] Candler T, Murphy R, Pigott A, Gregory JW. Fifteen-minute consultation: Diabulimia and disordered eating in childhood diabetes. Arch Dis Child Educ Pract Ed. 2018 Jun;103(3):118-123. doi: 10.1136/archdischild-2017-312689. Epub 2017 Oct 27. PMID 29079591
- [Background] Young V, Eiser C, Johnson B, Brierley S, Epton T, Elliott J, Heller S. Eating problems in adolescents with Type 1 diabetes: a systematic review with meta-analysis. Diabet Med. 2013 Feb;30(2):189-98. doi: 10.1111/j.1464-5491.2012.03771.x. PMID 22913589
- [Background] Winkley K, Ismail K, Landau S, Eisler I. Psychological interventions to improve glycaemic control in patients with type 1 diabetes: systematic review and meta-analysis of randomised controlled trials. BMJ. 2006 Jul 8;333(7558):65. doi: 10.1136/bmj.38874.652569.55. Epub 2006 Jun 27. PMID 16803942
- [Background] Hilliard ME, Powell PW, Anderson BJ. Evidence-based behavioral interventions to promote diabetes management in children, adolescents, and families. Am Psychol. 2016 Oct;71(7):590-601. doi: 10.1037/a0040359. PMID 27690487
- [Background] Golan M, Crow S. Targeting parents exclusively in the treatment of childhood obesity: long-term results. Obes Res. 2004 Feb;12(2):357-61. doi: 10.1038/oby.2004.45. PMID 14981230
- [Background] Jewell T, Blessitt E, Stewart C, Simic M, Eisler I. Family Therapy for Child and Adolescent Eating Disorders: A Critical Review. Fam Process. 2016 Sep;55(3):577-94. doi: 10.1111/famp.12242. Epub 2016 Aug 19. PMID 27543373
- [Background] Geist R, Heinmaa M, Stephens D, Davis R, Katzman DK. Comparison of family therapy and family group psychoeducation in adolescents with anorexia nervosa. Can J Psychiatry. 2000 Mar;45(2):173-8. doi: 10.1177/070674370004500208. PMID 10742877
- [Background] Nicholls DE, Yi I. Early intervention in eating disorders: a parent group approach. Early Interv Psychiatry. 2012 Nov;6(4):357-67. doi: 10.1111/j.1751-7893.2012.00373.x. Epub 2012 Jul 3. PMID 22759660
- [Background] Scott S. National dissemination of effective parenting programmes to improve child outcomes. Br J Psychiatry. 2010 Jan;196(1):1-3. doi: 10.1192/bjp.bp.109.067728. PMID 20044650
- [Background] Couturier J, Kimber M, Szatmari P. Efficacy of family-based treatment for adolescents with eating disorders: a systematic review and meta-analysis. Int J Eat Disord. 2013 Jan;46(1):3-11. doi: 10.1002/eat.22042. Epub 2012 Jul 23. PMID 22821753
- [Background] Hart LM, Damiano SR, Chittleborough P, Paxton SJ, Jorm AF. Parenting to prevent body dissatisfaction and unhealthy eating patterns in preschool children: a Delphi consensus study. Body Image. 2014 Sep;11(4):418-25. doi: 10.1016/j.bodyim.2014.06.010. Epub 2014 Aug 9. PMID 25084034
- [Background] Markowitz JT, Butler DA, Volkening LK, Antisdel JE, Anderson BJ, Laffel LM. Brief screening tool for disordered eating in diabetes: internal consistency and external validity in a contemporary sample of pediatric patients with type 1 diabetes. Diabetes Care. 2010 Mar;33(3):495-500. doi: 10.2337/dc09-1890. Epub 2009 Dec 23. PMID 20032278
- [Background] Markowitz JT, Volkening LK, Butler DA, Antisdel-Lomaglio J, Anderson BJ, Laffel LM. Re-examining a measure of diabetes-related burden in parents of young people with Type 1 diabetes: the Problem Areas in Diabetes Survey - Parent Revised version (PAID-PR). Diabet Med. 2012 Apr;29(4):526-30. doi: 10.1111/j.1464-5491.2011.03434.x. PMID 21883443
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Eisler I, Lock J, Le Grange D. Family-based treatments for Adolescents with Anorexia Nervosa. In The treatment of eating disorders: A clinical handbook. 1st ed. Guildford Press; 2011.
- [Background] Lock J, Le Grange. Treatment Manual for Anorexia Nervosa. A Family-Based Approach. 2nd ed. Guildford Press; 2015.
- [Background] National Collaborating Centre for Mental Health (UK). Eating Disorders: Core Interventions in the Treatment and Management of Anorexia Nervosa, Bulimia Nervosa and Related Eating Disorders. Leicester (UK): British Psychological Society (UK); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK49304/ PMID 23346610
- [Background] National Collaborating Centre for Mental Health (2015). Access and Waiting Time Standard for Children and Young People with an Eating Disorder. Commissioning guide. (July). Available from: https://www.england.nhs.uk/wp-content/uploads/2015/07/cyp-eating-disorders-access-waiting-timestandardcomm-guid.pdf
- [Background] Treasure J, Smith G, Crane A. Skills-based learning for caring for loved one with an eating disorder. 1st ed. Routledge; 2007.
- [Background] Andrews S, Charig R, Hale L, Draycott S. Evaluation of a psychoeducation group for parents with a young person with an eating: prelimary findings. Poster presentation at the International Eating Disorder Conference, London; 2019.
- [Background] Akhter K, Turnbull T, Simmons D. A systematic review of parent/peer-based group interventions for adolescents with type 1 diabetes: interventions based on theoretical/therapeutic frameworks. Br J Diabetes 2018;18:51-65.
- [Derived] Jones CJ, O'Donnell N, John M, Cooke D, Stewart R, Hale L, Skene SS, Kanumakala S, Harrington M, Satherley RM. PaRent InterventiOn to pRevent dIsordered eating in children with TYpe 1 diabetes (PRIORITY): Study protocol for a feasibility randomised controlled trial. Diabet Med. 2022 Apr;39(4):e14738. doi: 10.1111/dme.14738. Epub 2021 Nov 12. PMID 34741779